CLINICAL TRIAL: NCT00035802
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled 4-Week Study of the Safety and Efficacy of Topiramate in Adolescents With Acute Manic or Mixed Episodes of Bipolar I Disorder, With an Optional 6-Month Open-Label Extension
Brief Title: A Study to Evaluate the Safety and Effectiveness of Topiramate Compared to Placebo in the Treatment of Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: SR DIRECTOR CLINICAL LEADER, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016867; TOPMAT-PDMD-009
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Bipolar Disorder; Affective Disorders, Psychotic; Mood Disorders; Mental Disorders
Keywords: Bipolar; Mania; Pediatric; Children; Adolescent; Topiramate; Anticonvulsants; Central Nervous System Agents; Protective Agents; Neuroprotectiive Agents
MeSH Terms: conditions — Bipolar Disorder; Affective Disorders, Psychotic; Mood Disorders; Mental Disorders; Mania | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 001 (Experimental): Topiramate Double-blind period: Up to 400 mg/day (two 100-mg tablets twice a day) for 28 days.
  OL period: Up to 600 mg/day (three 100-mg tablets twice a day) for at least 6 months.
  Interventions: Drug: Topiramate
- 002 (Placebo Comparator): Placebo Double-blind period: Equal number of matching placebo tablets for each of the topiramate tablet strengths twice a day for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Double-blind period: Up to 400 mg/day (two 100-mg tablets twice a day) for 28 days.
  OL period: Up to 600 mg/day (three 100-mg tablets twice a day) for at least 6 months.
  Arms: 001
Drug: Placebo — Double-blind period: Equal number of matching placebo tablets for each of the topiramate tablet strengths twice a day for 28 days.
  Arms: 002

SUMMARY:
The purpose of this study is to determine the safety and efficacy of topiramate in adolescents with manic or mixed episodes of Bipolar I Disorder.

DETAILED DESCRIPTION:
This is a 4-week study to evaluate the safety and effectiveness of topiramate compared to placebo in the treatment of Bipolar I Disorder with an optional 6-month open-label (OL) extension for qualified patients following completion of the study. On Days 1-28 patients will receive placebo or topiramate 2x/day by mouth except for the 1st and last doses which will be a single evening dose and a single morning dose, respectively. Study drug will be titrated in 100-mg increments to 400 mg/day and patients maintained on a stable dose through Day 28. During the OL extension phase, topiramate will be titrated over 5 days to 200 mg/day. After Day 7, topiramate may be tapered down to 100 mg/day or up to 600 mg/day, as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Bipolar I Disorder (confirmed by the Kiddie-Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version [K-SADS-P/L])
* YMRS score greater than or equal to 20
* General good health as determined by medical history, physical examination, and laboratory evaluations
* Ability to swallow tablets
* Patient's parent or guardian must be fully capable of monitoring the patient's disease process and compliance to treatment
* Parent(s) or legal guardian(s) must read and sign the informed consent form after the nature of the study has been fully explained and assent must be obtained from patients

Exclusion Criteria:

* DSM-IV Axis I disorder diagnoses of autistic disorder, schizophrenia, schizoaffective disorder, or other psychotic disorders not otherwise specified (NOS)
* DSM-IV diagnosis of alcohol or substance dependence, with the exception of nicotine or caffeine dependence, within the 3 months prior to baseline. Acute or intermittent substance abuse prior to screening will not be exclusionary, depending upon the clinical judgment of the investigator
* Chronic antidepressant treatment within 4 weeks of randomization (5 weeks for fluoxetine), use of psychostimulants in the 7 days prior to baseline, use of any other psychotropic medications within 3 days or 5 half-lives, whichever is less, prior to baseline, or requirement for treatment with other psychotropic drugs on an ongoing basis
* Weight less than 33 kg or current or past history of anorexia nervosa
* Serious or unstable medical or neurological conditions

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2002-01; Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total Young Mania Rating Scale (YMRS) score | Baseline to Day 28 (or last available observation prior to Day 28).

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression Scale (CGI-S) score | Baseline to Day 28 (or last available observation prior to Day 28).
Change from baseline in Children's Global Assessment Scale (C-GAS) score | Baseline to Day 28 (or last available observation prior to Day 28).
The number of patients continuing to meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for manic or mixed episodes of Bipolar I Disorder | Day 28 (or last available observation prior to Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.